CLINICAL TRIAL: NCT06976372
Title: A Phase 1, Randomized, Double-blind, Multiple-dose Study to Evaluate the Pharmacokinetics of AMG 133 Administered Subcutaneously in Subjects With Overweight or Obesity
Brief Title: A Study to Evaluate AMG 133 Administered Subcutaneously in Participants With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 20240195
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Maridebart cafraglutide; AMG 133
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AMG 133 Dose A (Experimental): Participants will receive AMG 133 Dose A SC, followed by subsequent doses of Dose C and Dose D.
  Interventions: Drug: AMG 133
- AMG 133 Dose B (Experimental): Participants will receive AMG 133 Dose B SC, followed by subsequent doses of Dose C and Dose D.
  Interventions: Drug: AMG 133
- AMG 133 Dose C (Experimental): Participants will receive AMG 133 Dose C SC, followed by subsequent doses of Dose C and Dose D.
  Interventions: Drug: AMG 133

INTERVENTIONS:
Drug: AMG 133 — AMG 133 will be administered SC. Dose levels range from A to D lowest to highest.

SUMMARY:
The primary objective of this study is to assess the pharmacokinetics (PK) of AMG 133 after multiple subcutaneous (SC) administrations in participants with overweight or obesity using various dose regimens.

ELIGIBILITY:
Inclusion Criteria

1. Participant has provided informed consent before initiation of any study-specific activities/procedures.
2. Male or female participants, between 18 and 65 years of age (inclusive) at the time of Screening.
3. Except for obesity, no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [e.g., suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) as assessed by the Investigator (or designee). Participants with obstructive sleep apnea, controlled hypertension, and/or controlled dyslipidemia on stable therapies will be permitted. Participants with other mild, well-controlled comorbidities may be permitted with approval of the Investigator (or designee) in consultation with the Medical Monitor as appropriate.
4. Body mass index ≥ 27 kg/m^2 at the time of Screening.
5. Have a stable body weight (< 5 kg self-reported change) within 3 months before Screening, as assessed by the Investigator (or designee) based on participant self-report. Have not modified diet or adopted any nutritional lifestyle modification for 3 months, as assessed by the Investigator (or designee) based on participant self-report.

Exclusion Criteria

1. History or evidence, at Screening or Check-in, of clinically significant disorder, condition, or disease not otherwise excluded that, in the opinion of the Investigator (or designee), would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.
2. History of or active diabetes (regardless of type with the exception of gestational diabetes), or Hemoglobin A1C ≥ 6.5% (≥ 48 mmol/mol), at Screening.
3. History or evidence of endocrine disorder (such as Cushing's Syndrome) that can cause obesity.
4. History of acute or chronic pancreatitis within 1 year prior to Check-in, or elevation in serum lipase/amylase (> 2x the upper limit of normal) at Screening, or fasting serum triglyceride level of > 500 mg/dL at Screening. One repeat of abnormal values will be allowed.
5. Malignancy except nonmelanoma skin cancers or cervical or breast ductal carcinoma in situ within the last 5 years.
6. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2.
7. Uncontrolled thyroid disease, defined as thyroid-stimulating hormone (TSH) > 6.0 mIU/L or < 0.4 mIU/L at Screening. Participants who receive treatment for hypothyroidism are permitted if their thyroid hormone replacement dose has been stable for 3 months prior to Screening and TSH criteria are met.
8. History of or current signs of gastroparesis.
9. Previous surgical procedure for obesity within 6 months prior to Check-in.
10. History or current signs or symptoms of cardiovascular disease (aside from controlled hypertension and controlled dyslipidemia), including but not limited to myocardial infarction, congenital heart disease, valvular heart disease, coronary revascularization, or angina.
11. History or evidence of clinically significant arrhythmia at Screening, including any clinically significant findings on the ECG taken at Screening or Check-in.
12. History of hypersensitivity or allergy to AMG 133 or its ingredients, unless approved by the Investigator (or designee) and in consultation with the Sponsor.
13. Estimated glomerular filtration rate less than ≤ 60 mL/min/1.73 m^2 as calculated by the Modification of Diet in Renal Disease equation at Screening or Check-in. One repeat of abnormal values will be allowed.
14. Alanine aminotransferase or aspartate aminotransferase > 2x the upper limit of normal at Screening or Check-in. One repeat of abnormal values will be allowed.
15. History of or current suicidal ideation (thoughts), suicide attempt(s), or major psychiatric illness (including depression) within 6 months prior to Screening.
16. Use of any over-the-counter or prescription medications within 30 days or 5 half-lives (whichever is longer) before Check-in.
17. Current use or prior use of any glucagon-like peptide 1 receptor (GLP-1R) agonist, GIPR glucose-dependent insulinotropic polypeptide receptor (GIPR) agonist or antagonist within the past 3 months prior to Check-in.
18. Current or prior use of all herbal medicines (e.g., St. John's wort), vitamins, and supplements consumed by the participant within the 30 days prior to enrollment, unless deemed acceptable by the Investigator (or designee) and in consultation with the Sponsor.
19. Female participants of childbearing potential with a positive pregnancy test assessed at Screening or Check-in by a serum or urine pregnancy test.
20. Female participants lactating/breastfeeding or who plan to breastfeed during the study through 16 weeks after the last dose of AMG 133.
21. Unwilling to adhere to contraceptive requirements through 16 weeks after the last dose of AMG 133.
22. Participant has received a dose of an investigational drug within the past 30 days or 5 half-lives, whichever is longer, prior to Check-in.
23. Have previously completed or withdrawn from this study or any other study investigating AMG 133 or have previously received the investigational product.
24. Unwilling to abide with study restrictions.
25. Participants who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Maximum Concentration (Cmax) of AMG 133 | Up to Day 99
Area Under the Plasma Concentration-time Curve from Time Zero to the Last Quantifiable Concentration (AUClast) of AMG 133 | Day 29
Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUCinf) of AMG 133 | Day 29
Area Under the Plasma Concentration-time Curve Over the Dosing Interval (AUCtau) of AMG 133 | Day 1 and Day 15

SECONDARY OUTCOMES:
Number of Participants Who Experience Treatment-emergent Adverse Events | Up to Day 99
Number of Participants Who Experience Serious Adverse Events | Up to Day 99
Number of Participants Who Develop Anti-AMG 133 Antibodies | Up to Day 99

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - CenExel, Anaheim, California
  - CenExel Collaborative Neuroscience Research, LLC Los Alamitos, Los Alamitos, California
  - Fortrea Clinical Research Unit - Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com